CLINICAL TRIAL: NCT03273816
Title: Evaluation of the Benefit Provided by Sessions of Sophrology on the Intraoperative Management of Parkinsonian Patients in the Context of Deep Brain Stimulation Surgery.
Brief Title: Evaluation of the Benefit Provided by Sessions of Sophrology on the Per Operative Management of Parkinsonian Patients Planned for a Deep Brain Stimulation Surgery.
Acronym: SOPHROSTIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment rate
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35RC16_9805
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, bi-centric (national), superiority, open-label, blind-blind (evaluator) trial comparing sophrology to routine care in preparation for deep brain stimulation. The distribution of patients will be balanced between the two groups.
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint is taken by a nurse who does not know the randomization arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without sessions of sophrology (No Intervention): The control group is also composed of Parkinsonian patients waiting for deep brain surgery but will not have any special preparation for the procedure. They will be subjected to the same assessments at the same time as the sophrology group.
- Patients with sessions of sophrology (Experimental): The experimental group is composed of patients with Parkinson's waiting for deep brain surgery. They will benefit from 10 sessions of sophrology in preparation for the intervention 5 weeks before this one.
  Interventions: Behavioral: sessions of sophrology

INTERVENTIONS:
Behavioral: sessions of sophrology — 10 sessions of sophrology in preparation for the intervention 5 weeks before this one.
  Arms: Patients with sessions of sophrology

SUMMARY:
Deep brain stimulation surgery, which consists of intracerebral implantation of electrodes, is considered one of the most effective techniques for controlling the motor fluctuations of Parkinson's disease. The particularity of this surgery is the necessity of the awakening of the patient for the correct positioning of the electrodes, it is therefore a difficult test for the patient.

Medical sophrology is an ideal strategy to optimize the comfort of the patient during the operation thanks to its anxiolytic and analgesic virtues while guaranteeing the maintenance of a good patient vigilance favoring the cooperation with the operating room team. Indeed, sophrology is a body-mediated set of techniques, at the crossroads between hypnosis and yoga, which makes it possible to find a balance between emotions, thoughts and behaviors. It has already been applied in other fields such as oncology, pain management, preparation for childbirth, and for 5 years at the CHU of Rennes for preparation for the intervention of deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age greater than or equal to 18 years)
* Patient with idiopathic Parkinson's disease with programmed deep brain stimulation (VIM target, NST, single or bilateral GPI);
* Planned intervention in an awake patient (implying MOCA> 21 (Montreal Cognitive Assessment));
* Patient understanding the course of the study;
* Patient who has given informed consent in writing;
* Patient benefiting from a system of social insurance.

Exclusion Criteria:

* - Intervention under general anesthesia;
* Pregnant or nursing women;
* Major person under protective measures (safeguard of justice, curatorship and guardianship);
* Person deprived of liberty.
* Patient having already had a practice in yoga, sophrology, hypnotherapy superior or equal to 5 sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Patient anxiety | at one hour after the beginning of the intervention
  patient anxiety evaluated by the STAI-YA (State Trait Anxiety Inventory), retranscribed by a caregiver of the block, the patient being unable in practice to fill in a questionnaire at that time

SECONDARY OUTCOMES:
Per operative pain | intraoperative (at the beginning of the intervention)
  Per operative pain judged by a visual scale analogous
Per operative pain | at one hour after the begginnig of the intervention
  Per operative pain judged by a visual scale analogous
Per operative pain | Intraoperative (At the end of the first electrode placement)
  Per operative pain judged by a visual scale analogous
Evaluation of the anxiety | At one hour before the procedure
  Evaluation of the anxiety measured by the STAI YA
Evaluation of the anxiety | Intraoperative (At the end of the first electrode placement)
  Evaluation of the anxiety measured by the STAI YA
Interaction between the patient and the surgical team during the procedure | At Day 0
  interaction is judged by a visual analogue scale to be completed by the neurologist and the neurosurgeon
The duration of the intervention in minutes | intraoperative
  The duration of the intervention in minutes
Heart rate | At one hour after the beginning of the intervention
  Heart rate in beat per minute
Blood pressure | At one hour after the beginning of the intervention
  Blood pressure in mmHg
Experience of the surgical intervention | At 24 hours after surgery
  experience of the surgical intervention by the patient evaluated on a visual analog scale
Experience of the surgical intervention | one week after surgery
  experience of the surgical intervention by the patient evaluated on a visual analog scale
Experience of the perioperative period by the patient | one week after surgery
  Qualitative analysis
Occurrence adverse event | Through study completion (Day 0 to Week 1)
  Occurrence of hematoma
Occurrence adverse event | Through study completion (Day 0 to Week 1)
  Occurrence of infection
Occurrence adverse event | Through study completion (Day 0 to Week 1)
  Occurrence of dysfunction of material
Inter-group comparison of the evolution of anxiety | between the inclusion (Month -3) and the beginning of the intervention (Hour O)
  Inter-group comparison of the evolution of anxiety by the STAI-YA

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERIN, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided